CLINICAL TRIAL: NCT05639075
Title: Effect of an Intraocular Lens With Enhanced Peripheral Vision on Gait Performance: a Pilot Study
Brief Title: Analysis of Peripheral Vision With Two Different IOLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Voptica
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Cataract
Keywords: Cataract; Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait analysis (Experimental): A gait analysis test will be performed in each patient after cataract surgery to test peripheral vision
  Interventions: Other: Peripheral vision

INTERVENTIONS:
Other: Peripheral vision — A gait analysis test will be performed in each patient after cataract surgery to test peripheral vision

SUMMARY:
Analyse the peripheral vision after cataract surgery with a new IOL compared to a standard IOL

DETAILED DESCRIPTION:
Due to continuous improvements in the technique of cataract surgery as well as the material and the design of the intraocular lenses (IOLs) over the few past decades, the removal of the opacified lens is considered to be relatively safe surgery with good refractive outcomes and a short rehabilitation time. In conjunction with these improvements of the procedure, the patients' expectations concerning their postoperative visual quality and refractive outcomes are increasing.

Different IOLs have been developed to satisfy the patients' demands. Standard monofocal IOL offer good vision in either the far or the near distance, whereas spectacles are still needed for all other distances. On the other hand, multifocal IOLs allow freedom of glasses in all of the three distances (far, intermediate, near), but are, in most cases, associated with a decrease in contrast sensitivity and induction of disturbing photic phenomena (e.g., halo, starbursts, glare).

Enhanced depth of focus (EDOF) IOLs are another lens option and promise good intermediate vision combined with good vision in the far distance, with spectacles only being needed for reading tasks. However, like multifocal IOLs, these lenses may be accompanied by photic phenomena, although to a lesser extent than with multifocal IOL. Recently, the so-called enhanced monofocal IOLs were introduced to the market. These IOLs are comparable to other monofocal IOLs concerning contrast sensitivity and photic phenomena, but besides offering good far visual acuity, they also slightly enhance the depth of focus with some intermediate distance vision.

However, all of these lenses only provide optimal image quality in the very central visual field. Indeed it was shown that in pseudophakic patients the peripheral vision is decreased compared to phakic patients, reducing the peripheral image quality compared to that of the natural crystalline lens. According to computational and physical modelling experiments, this effect may be due to a higher degree of astigmatism and increased higher-order aberrations (HOAs) in the IOL periphery compared to those of the natural lens. This increase in astigmatism was observed in all pseudophakic individuals and did not depend on the power or the type of the implanted IOL. Peripheral vision is thought to have an impact on contrast resolution and sensitivity, detection of small stimuli and the movement of targets in the periphery, exploration and interpretation of a scene, and peripheral visual crowding. All of these tasks are important for the orientation and navigation of patients in their everyday life and misinterpretation of a scene or missing details while walking may lead to an increased risk of falls or accidents. Therefore, an IOL that improves peripheral vision could lead to a better overall functional visual quality and even patients with loss of central vision might benefit from such devices.

Recently, a new non-diffractive inverted meniscus EDOF IOL, the Art40 IOL, which reduces peripheral astigmatism was introduced to the market. This IOL promises to mimic the natural crystalline lens leading to optimized field curvature, improvement in peripheral vision, and enhanced contrast sensitivity of the patients without introducing photic phenomena. Therefore, the aim of this study is to analyse if the peripheral vision after cataract surgery is increased in patients with this new IOL compared to a standard IOL.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic patients with an Art 40 IOL in one eye and the standard monofocal ICB00 IOL in the other eye. A larger series of patients was operated in this way at Hanusch hospital in 2021 and 2022 as the department has the strategy of implanting a new IOL that has come to market in only one eye and the standard monofocal IOL in the contralateral eye to reduce potential risks, even though the new IOL had a CE mark and was readily available on the market.
* Surgery should have been at least 1 month prior to study recruitment
* Age 21 or older
* Visual acuity > 0,8
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Able to walk without walking aids
* Written informed consent prior to commencing study measurements.

Exclusion Criteria:

* nystagmus or pathologies that might affect patient's fixation or physical handicaps that may decrease gait stability
* any ophthalmic comorbidity that may compromise the visual function or might interfere with the experiments (e.g., macular degeneration, corneal scars, pupil abnormalities, glaucoma)
* reduced contrast sensitivity, binocularity, and stereoscopic vision (e.g., amblyopia, strabismus)
* limitation of age-equivalent gait performance because of neurological, cardio-respiratory or musculoskeletal functional deficits
* pregnancy (pregnancy test will be performed in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral vision | 24 months
  Peripheral vision will be assessed via gait analysis and will be compared between both eyes

SECONDARY OUTCOMES:
Refraction | 24 months
  Refraction will be assessed with trial frames and will be compared between both eyes
Visual acuity | 24 months
  Visual acuity will be assessed with ETDRS charts and will be compared between both eyes

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided